CLINICAL TRIAL: NCT02871193
Title: Study of Ultrasound-guided Thoracic Paravertebral Block Using Ropivacaine With/Without Dexamethasone in Elective Thoracotomy
Brief Title: Ultrasound-guided Thoracic Paravertebral Block Using Ropivacaine With/Without Dexamethasone in Elective Thoracotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Kuai2016-06-08
Record Dates: First submitted 2016-07-17; First posted 2016-08-18 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Surgery
Keywords: paravertebral block; patient controlled analgesia; ropivacaine; dexamethasone
MeSH Terms: interventions — Ropivacaine; Dexamethasone; Calcium Dobesilate; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group C（Control） (Sham Comparator): Group C received ultrasound-guided thoracic paravertebral nerve block (TPVB) with 0.9% saline 20ml combined with general anesthesia and intravenous patient controlled analgesia pump.
  Interventions: Other: saline
- Group R(Ropivacaine) (Experimental): Group R received ultrasound-guided thoracic paravertebral nerve block (TPVB) with 0.5% ropivacaine 20 ml combined with general anesthesia and intravenous patient controlled analgesia pump.
  Interventions: Drug: Ropivacaine
- Group D(Dexamethasone) (Experimental): Group D received ultrasound-guided thoracic paravertebral nerve block (TPVB) with 0.5% ropivacaine 20ml and dexamethasone 5 mg combined with general anesthesia and intravenous patient controlled analgesia pump.
  Interventions: Drug: Ropivacaine; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ropivacaine — ultrasound-guided thoracic paravertebral nerve block (TPVB) with 0.5% ropivacaine 20ml
  Other Names: ropivacaine hydrochloride
  Arms: Group D(Dexamethasone); Group R(Ropivacaine)
Drug: Dexamethasone — ultrasound-guided thoracic paravertebral nerve block (TPVB) with 0.5% ropivacaine 20ml and dexamethasone 5 mg
  Other Names: dxm; dex
  Arms: Group D(Dexamethasone)
Other: saline — ultrasound-guided thoracic paravertebral nerve block (TPVB) with 0.9% saline 20ml
  Other Names: normal saline
  Arms: Group C（Control）

SUMMARY:
The procedures of thoracotomy are among the most painful operations. In addition to post-thoracotomy pain, the outcomes of surgery are affected adversely by postoperative discomfort. Therefore, post-thoracotomy pain control can improve the satisfaction of patient and prevent postoperative complications such as pneumonia, atelectasis, or respiratory failure. Thoracic epidural analgesia (TEA) used to be widely considered as a standard technique for providing analgesia after a thoracotomy. However, TEA carries side-effects such as incomplete or failed block, epidural hematoma, abscess, hypotension, respiratory depression, or bradycardia, etc. Recently, thoracic paravertebral block (TPVB) is an alternative technique for TEA that may offer a comparable analgesic effect and a better side -effect profile for post-thoracotomy analgesia. When local anesthetic agents are used as single injection, they can provide analgesia for limited period. Various adjuvants have been tried in the past in order to enhance the duration and quality of postoperative analgesia. Previous studies with perineural dexamethasone demonstrated that it enhanced the duration of local anesthetic block. The mechanism of its action is blocking the nociceptive impulse transmission along the myelinated C fibers. Patient-controlled analgesia (PCA) devices have been shown to provide superior analgesia and greater patient satisfaction compared with intermittent administration. System of wire-less PCA provides remote monitoring, information management and PCA devices with high precision. The purpose of this research is to determine whether dexamethasone might prolong the duration of analgesia and improve the short-time outcomes when administered for TPVB along with local anesthetic agents in elective thoracotomy.

ELIGIBILITY:
Inclusion Criteria:

1. patient American Society of Anesthesiologists（ASA） I~III undergoing elective thoracotomy
2. written informed consent from the patient or the relatives of the participating patient

Exclusion Criteria:

1. mental illness
2. thoracic paravertebral blocks contraindicated
3. local anesthetic allergy
4. people who have heart disease
5. people who have severe liver or renal disease
6. people who have severe endocrine disease
7. people who can't communicate effectively because of hearing or visual disorders

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2016-10-08 (Actual); Study Completion 2017-01-20 (Actual)

PRIMARY OUTCOMES:
the change of visual analogue scale(VAS) of patients with different treatment-related events in the following 3 days after thoracotomy | 6 hours,12hours,24hours and 72hours after operation
  to show the grading of pain in different groups after surgery
the reality pressing number of patient controlled analgesia(PCA) of patients with different treatment-related events in the following 3 days after surgery | 6hours,12hours,24hours and 72hours after operation
  to show the consumption of analgesics after surgery

SECONDARY OUTCOMES:
hemodynamic index | 24 hours after anesthesia
  To show the changing trend of hemodynamics with different treatment-related events when receiving thoracotomy.
The time of recovery | 24 hours after surgery
  to show the quality of recovery
The time of extubation | 24 hours after surgery
  to show the quality of recovery
the incidence of side effects | 3days after operation
  To compare the incidence rates of side effects, such as nausea, vomiting, dizziness, hypotension and bradyarrhythmia in the first 3 days after operation.
The complication after surgery | 30 days after surgery
  To compare the incidence rates of complications, such as pneumonia, atelectasis, respiratory failure, heart failure, etc
The first day of leaving bed after surgery | 30 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of Anhui Medical University, Hefei, Anhui, China

REFERENCES:
- [Result] Carmona P, Llagunes J, Canovas S, de Andres J, Marques I. The role of continuous thoracic paravertebral block for fast-track anesthesia after cardiac surgery via thoracotomy. J Cardiothorac Vasc Anesth. 2011 Feb;25(1):205-6. doi: 10.1053/j.jvca.2010.04.005. No abstract available. PMID 20599397
- [Result] Tomar GS, Ganguly S, Cherian G. Effect of Perineural Dexamethasone With Bupivacaine in Single Space Paravertebral Block for Postoperative Analgesia in Elective Nephrectomy Cases: A Double-Blind Placebo-Controlled Trial. Am J Ther. 2017 Nov/Dec;24(6):e713-e717. doi: 10.1097/MJT.0000000000000405. PMID 26938764
- [Result] Ilfeld BM, Madison SJ, Suresh PJ, Sandhu NS, Kormylo NJ, Malhotra N, Loland VJ, Wallace MS, Proudfoot JA, Morgan AC, Wen CH, Wallace AM. Treatment of postmastectomy pain with ambulatory continuous paravertebral nerve blocks: a randomized, triple-masked, placebo-controlled study. Reg Anesth Pain Med. 2014 Mar-Apr;39(2):89-96. doi: 10.1097/AAP.0000000000000035. PMID 24448512
- [Result] Ke JD, Hou HJ, Wang M, Zhang YJ. The comparison of anesthesia effect of lung surgery through video-assisted thoracic surgery: A meta-analysis. J Cancer Res Ther. 2015 Nov;11 Suppl:C265-70. doi: 10.4103/0973-1482.170534. PMID 26612450
- [Result] Albrecht E, Kern C, Kirkham KR. A systematic review and meta-analysis of perineural dexamethasone for peripheral nerve blocks. Anaesthesia. 2015 Jan;70(1):71-83. doi: 10.1111/anae.12823. Epub 2014 Aug 14. PMID 25123271